CLINICAL TRIAL: NCT04288674
Title: Leptospirosis Registry - LeptoScope
Acronym: Leptoscope
Status: Recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, Principal Investigator, University of Cologne
Other Study IDs: Version 1.0
Record Dates: First submitted 2020-02-12; First posted 2020-02-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Leptospirosis
MeSH Terms: conditions — Leptospirosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Leptospirosis group: Patients with cultural, serological, molecular or histological evidence and clinical evidence of invasive leptospirosis disease.
  Interventions: Other: Retrospective data collection of demographics; Other: Retrospective data collection of underlying diseases; Other: Retrospective data collection of duration of hospitalization
- Control group: Controls will be included at the same hospitals that conduced cases based on matching of demographics, underlying diseases and duration of hospitalization (i.e. one control per case, both in the same hospital)
  Interventions: Other: Retrospective data collection of demographics; Other: Retrospective data collection of underlying diseases; Other: Retrospective data collection of duration of hospitalization

INTERVENTIONS:
Other: Retrospective data collection of demographics — Retrospective data collection of demographics from patients with leptospirosis and matching control group patients.
Other: Retrospective data collection of underlying diseases — Retrospective data collection of underlying diseases from patients with leptospirosis and matching control group patients.
Other: Retrospective data collection of duration of hospitalization — Retrospective data collection of duration of hospitalization from patients with leptospirosis and matching control group patients.

SUMMARY:
Leptospirosis is a worldwide zoonotic diseases caused by pathogenic Leptospira spp. Human are accidental hosts, who acquired infections after exposition to animal urine, contaminated water or soil, infected tissue. Incidence of invasive leptospirosis disease causing acute kidney injury, acute respiratory distress syndrome (ARDS), myocarditis, hepatic dysfunction, hemorrhage and multi-organ failure, is globally increasing and there have been frequent outbreak situation throughout the world. Due to increasing outbreak situations and globally chances in species distributions, a worldwide surveillance in epidemiology and species distribution is urgently needed. The objective of the Leptospirosis Registry - LeptoScope is to overcome the lack knowledge on epidemiology, clinical course, prognostic factors and molecular characteristics for invasive leptospirosis disease.

DETAILED DESCRIPTION:
Leptospirosis is a worldwide zoonotic diseases caused by pathogenic Leptospira spp. Human are accidental hosts, who acquired infections after exposition to animal urine, contaminated water or soil, infected tissue. During bacteremia, Leptospira spp. may lead to invasive, deep-seated leptospirosis with infection of kidney, liver, heart and the central nervous system. Although cleaned from blood and most tissue by immune response, Leptospira spp. can persists and multiply in the tubuli of kidneys.

Incidence of invasive leptospirosis disease causing acute kidney injury, acute respiratory distress syndrome (ARDS), myocarditis, hepatic dysfunction, hemorrhage and multi-organ failure, is globally increasing and there have been frequent outbreak situation throughout the world. In Europe, invasive leptospirosis disease is less common than in the tropical and subtropical countries, however due to climate change incidence is rising, and there are worry-some trends concerning chancing species distribution and multiple outbreak situations throughout central Europe. Current treatment approaches consist of antibiotic therapies. Additionally, salvage supportive treatment approaches of critical ill patients are common in invasive leptospirosis disease requiring dialysis, hemodynamic support, mechanical ventilation or even extracorporeal membrane oxygenation (ECMO). Furthermore, invasive leptospirosis disease is associated with the development of chronic kidney disease.

Due to increasing outbreak situations and globally chances in species distributions, a worldwide surveillance in epidemiology and species distribution is urgently needed. Additionally, the examination of attributable mortality and costs analysis of invasive leptospirosis disease will need to be studied on a multinational basis and therefore LeptoScope will particularly use a matched case control design.

The objective of the Leptospirosis Registry - LeptoScope is to overcome the lack knowledge on epidemiology, clinical course, prognostic factors and molecular characteristics for invasive leptospirosis disease. Additionally, LeptoScope serves as a platform for monitoring complications of invasive leptospirosis disease and outbreak situations.

ELIGIBILITY:
Inclusion Criteria:

* Cultural, serological, molecular or histological evidence of invasive leptospirosis diseases
* Clinical signs of disseminated leptospirosis disease without cultural, serological, molecular or histological evidence
* Case controls: Matching procedures for controls: Particularly, case controls will be included at the same hospitals that conduced cases based on matching of demographics, underlying diseases and duration of hospitalization (i.e. one control per case, both in the same hospital).

Exclusion Criteria:

* Colonization or other non-invasive infection
* Cultural, serological, molecular or histological evidence without dissemination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective data collection from patients with cultural, serological, molecular or histological evidence of Leptospirosis spp. infection and clinical evidence of invasive leptospirosis disease (acute kidney injury, pulmonary manifestation with acute respiratory distress syndrome (ARDS), myocarditis with arrhythmia, hepatic dysfunction, hemorrhage, multi-organ failure).
  Particularly, controls will be included at the same hospitals that conduced cases based on matching of demographics, underlying diseases and duration of hospitalization (i.e. one control per case, both in the same hospital).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence | up to 100 weeks
  To describe the global incidence of invasive leptospirosis disease
Mortality | up to 100 weeks
  To describe global mortality due to invasive leptospirosis disease

SECONDARY OUTCOMES:
Resistance development | up to 100 weeks
  To describe resistance developments of Leptospirosis spp.
Treatment efficacy of invasive leptospirosis disease in participants with treatment failure | at 90 days from diagnosis
  To describe the number of participants with treatment failure
Treatment efficacy of invasive leptospirosis disease in participants with stable disease | at 90 days from diagnosis
  To describe the number of participants with stable disease
Treatment efficacy of invasive leptospirosis disease in participants with partial responses | at 90 days from diagnosis
  To describe the number of participants with partial responses
Treatment efficacy of invasive leptospirosis disease in participants with complete responses | at 90 days from diagnosis
  To describe the number of participants with complete responses
Occurrence of acute kidney injury according to KDIGO I, II, III | at 90 days from diagnosis
  To describe the occurrence of acute kidney injury according to KDIGO I, II, III disease
Occurrence of chronic kidney disease | up to 500 weeks
  To describe the occurrence of chronic kidney disease
Need for renal replacement therapy | up to 500 weeks
  To describe the need for renal replacement therapy approaches

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Study Chair — University Hospital of Cologne; Felix Köhler, MD, Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related information — http://www.kidneyinfection.org/leptoscope/